CLINICAL TRIAL: NCT02185417
Title: CSP #597 - Diuretic Comparison Project
Brief Title: Diuretic Comparison Project
Acronym: DCP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 597
Record Dates: First submitted 2014-06-30; First posted 2014-07-09 (Estimated); Results first posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Hypertension
Keywords: Hypertension; Cardiovascular outcomes; Pragmatic clinical trial; Point of care research
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide; Chlorthalidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Hydrochlorothiazide (Active Comparator): Participants remained on the existing hydrochlorothiazide treatment regimen (a daily dose of 25 or 50 mg).
  Interventions: Drug: Hydrochlorothiazide (HCTZ)
- Chlorthalidone (Active Comparator): Participants switched to an equivalent dose of chlorthalidone (a daily dose of 12.5 or 25 mg).
  Interventions: Drug: Chlorthalidone (CTD)
- Providers (No Intervention): Providers were enrolled in order to contact their potentially eligible patients and were not included in the results

INTERVENTIONS:
Drug: Hydrochlorothiazide (HCTZ) — Trial activities following study randomization were considered as usual care. Prescriptions of the allocated drug were managed by the primary care providers and patients would receive the prescribed mediations through the VA outpatient pharmacy services.
  Other Names: HCTZ
  Arms: Hydrochlorothiazide
Drug: Chlorthalidone (CTD) — Trial activities following study randomization were considered as usual care. Prescriptions of the allocated drug were managed by the primary care providers and patients would receive the prescribed mediations through the VA outpatient pharmacy services.
  Other Names: CTD
  Arms: Chlorthalidone

SUMMARY:
The Diuretic Comparison Project aimed to evaluate whether chlorthalidone, as compared with hydrochlorothiazide, would reduce the risk of major nonfatal cardiovascular disease outcomes and non-cancer-related deaths in older patients with hypertension who were receiving hydrochlorothiazide at baseline. The investigators incorporated the pragmatic methods used by the Department of Veterans Affairs (VA) Healthcare System to provide a real-world assessment of the effectiveness of chlorthalidone as compared with hydrochlorothiazide in routine clinical care.

DETAILED DESCRIPTION:
Thiazide-type diuretics have been in use for more than 50 years and are considered as the first-line treatment for hypertension. Of the more than 1 million Veterans prescribed a thiazide-type diuretic each year, more than 95% receive hydrochlorothiazide, and fewer than 2.5% receive chlorthalidone. However, indirect evidence has been accumulating for many years that chlorthalidone may be more effective than hydrochlorothiazide at preventing cardiovascular events.

The Diuretic Comparison Project was conducted with a clinically integrated design (termed a "point of care" or "pragmatic embedded" trial). The key feature of our design was that, instead of employing local investigators, the investigators developed centralized trial procedures and implemented into the VA electronic health record (EHR) and healthcare delivery systems. This approach enabled us to conduct trial-related interactions and randomization with the use of data in the EHRs, centralize recruitment efforts without the use of site staff, eliminate the need for trial-related visits and procedures, and centralize data capture from administrative databases.

This study was performed to answer a question of whether chlorthalidone is more effective than hydrochlorothiazide at preventing cardiovascular outcomes. Consent was obtained from eligible participants who were willing to participate and their primary care providers. With provider assented to the patient undergoing randomization, 3,523 older patients with hypertension were randomized across 72 VA health care systems. Patients across the US (including Puerto Rico and District of Columbia) were enrolled. Participants were randomly assigned to continue with existing hydrochlorothiazide treatment regimen (25/50mg daily) or switch to a dose equivalent chlorthalidone (12.5/25 mg daily).

The primary outcome was the first occurrence of a composite outcome consisting of a nonfatal cardiovascular event or non-cancer related death. Nonfatal cardiovascular events included nonfatal myocardial infarction, stroke, hospitalization for heart failure, or urgent coronary revascularization for unstable angina.

ELIGIBILITY:
Inclusion criteria

* over age 65 years
* receiving hydrochlorothiazide from the VA pharmacy at a daily dose of 25 or 50 mg
* most recent SBP ≥120 mm Hg and no records of SBP <120 mm Hg in the past 90 days

Exclusion criteria:

* impaired decision-making capacity rendering the patient unable to provide informed consent (i.e., if there is any question during the nurse's EHR chart review that the individual does not have the ability to make an autonomous decision or the PCP declines permission to randomize)
* death expected within 6 months (inferred by PCP permission to randomize)
* blood potassium level <3.1 or 3.5 (if taking digoxin) meq/L in the past 90 days
* blood sodium level <130 meq/L in the past 90 days
* enrolled in Medicare Part C (This exclusion only applied if there might be insufficient EHR data available to the study team)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20723 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Areef Ishani, MD MS, Study Chair — Minneapolis VA Health Care System, Minneapolis, MN; William C Cushman, MD, Study Chair — Memphis VA Medical Center, Memphis, TN
Locations (68):
- United States (67):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - Alaska VA Healthcare System, Anchorage, AK, Anchorage, Alaska
  - Veterans Health Care System of the Ozarks, Fayetteville, AR, Fayetteville, Arkansas
  - Central Arkansas VHS John L. McClellan Memorial Veterans Hospital, Little Rock, AR, Little Rock, Arkansas
  - VA Central California Health Care System, Fresno, CA, Fresno, California
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - Grand Junction VA Medical Center, Grand Junction, CO, Grand Junction, Colorado
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Wilmington VA Medical Center, Wilmington, DE, Wilmington, Delaware
  - Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia
  - Bay Pines VA Healthcare System, Pay Pines, FL, Bay Pines, Florida
  - North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida
  - VA Pacific Islands Health Care System, Honolulu, HI, Honolulu, Hawaii
  - Boise VA Medical Center, Boise, ID, Boise, Idaho
  - VA Illiana Health Care System, Danville, IL, Danville, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - Captain James A. Lovell Federal Health Care Center, North Chicago, IL, North Chicago, Illinois
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - VA Central Iowa Health Care System, Des Moines, IA, Des Moines, Iowa
  - Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa
  - Maine VA Medical Center, Augusta, ME, Togus, Maine
  - Rehabilitation R&D Service, Baltimore, MD, Baltimore, Maryland
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Aleda E. Lutz VA Medical Center, Saginaw, MI, Saginaw, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - St. Cloud VA Health Care System, St. Cloud, MN, Saint Cloud, Minnesota
  - VA Gulf Coast Veterans Health Care System, Biloxi, MS, Biloxi, Mississippi
  - Kansas City VA Medical Center, Kansas City, MO, Kansas City, Missouri
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri
  - Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska
  - Manchester VA Medical Center, Manchester, NH, Manchester, New Hampshire
  - New Mexico VA Health Care System, Albuquerque, NM, Albuquerque, New Mexico
  - Albany VA Medical Center Samuel S. Stratton, Albany, NY, Albany, New York
  - Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York
  - Syracuse VA Medical Center, Syracuse, NY, Syracuse, New York
  - Durham VA Medical Center, Durham, NC, Durham, North Carolina
  - Fargo VA Healthcare System, Fargo, ND, Fargo, North Dakota
  - Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio
  - Dayton VA Medical Center, Dayton, OH, Dayton, Ohio
  - Jackson C. Montgomery VA Medical Center, Muskogee, OK, Muskogee, Oklahoma
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Roseburg Healthcare System, Roseburg, OR, Roseburg, Oregon
  - VA Southern Oregon Rehabilitation Center and Clinics, White City, OR, White City, Oregon
  - Coatesville VA Medical Center, Coatesville, PA, Coatesville, Pennsylvania
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - Wilkes-Barre VA Medical Center, Wilkes-Barre, PA, Wilkes-Barre, Pennsylvania
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - Wm. Jennings Bryan Dorn VA Medical Center, Columbia, SC, Columbia, South Carolina
  - VA Black Hills Health Care System Fort Meade Campus, Fort Meade, SD, Sturgis, South Dakota
  - Memphis VA Medical Center, Memphis, TN, Memphis, Tennessee
  - Tennessee Valley Healthcare System Nashville Campus, Nashville, TN, Nashville, Tennessee
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas
  - South Texas Health Care System, San Antonio, TX, San Antonio, Texas
  - White River Junction VA Medical Center, White River Junction, VT, White River Junction, Vermont
  - Hampton VA Medical Center, Hampton, VA, Hampton, Virginia
  - Huntington VA Medical Center, Huntington, WV, Huntington, West Virginia
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin
  - Clement J. Zablocki VA Medical Center, Milwaukee, WI, Milwaukee, Wisconsin
  - Tomah VA Medical Center, Tomah, WI, Tomah, Wisconsin
  - Sheridan VA Medical Center, Sheridan, WY, Sheridan, Wyoming
- VA Caribbean Healthcare System, San Juan, PR, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No
There is no IPD sharing plan description

REFERENCES:
- [Background] Ishani A, Leatherman SM, Woods P, Hau C, Klint A, Lew RA, Taylor AA, Glassman PA, Brophy MT, Fiore LD, Ferguson RE, Cushman WC. Design of a pragmatic clinical trial embedded in the Electronic Health Record: The VA's Diuretic Comparison Project. Contemp Clin Trials. 2022 May;116:106754. doi: 10.1016/j.cct.2022.106754. Epub 2022 Apr 4. PMID 35390512
- [Background] Ferguson RE, Leatherman SM, Woods P, Hau C, Lew R, Cushman WC, Brophy MT, Fiore L, Ishani A. Practical issues in pragmatic trials: the implementation of the Diuretic Comparison Project. Clin Trials. 2023 Jun;20(3):276-283. doi: 10.1177/17407745231160553. Epub 2023 Mar 29. PMID 36992530
- [Result] Ishani A, Cushman WC, Leatherman SM, Lew RA, Woods P, Glassman PA, Taylor AA, Hau C, Klint A, Huang GD, Brophy MT, Fiore LD, Ferguson RE; Diuretic Comparison Project Writing Group. Chlorthalidone vs. Hydrochlorothiazide for Hypertension-Cardiovascular Events. N Engl J Med. 2022 Dec 29;387(26):2401-2410. doi: 10.1056/NEJMoa2212270. Epub 2022 Dec 14. PMID 36516076
- [Result] Hau C, Efird JT, Leatherman SM, Soloviev OV, Glassman PA, Woods PA, Ishani A, Cushman WC, Ferguson RE. A Centralized EHR-Based Model for the Recruitment of Rural and Lower Socioeconomic Participants in Pragmatic Trials: A Secondary Analysis of the Diuretic Comparison Project. JAMA Netw Open. 2023 Sep 5;6(9):e2332049. doi: 10.1001/jamanetworkopen.2023.32049. PMID 37656456
- [Derived] Anand ST, Hau C, Davenport MJ, Ishani A, Cushman WC, Glassman PA, Taylor AA, Lew RA, Ferguson RE, Leatherman SM. Per-Protocol Analysis of Chlorthalidone Versus Hydrochlorothiazide for Cardiovascular Event Prevention-Diuretic Comparison Project. J Am Heart Assoc. 2026 Jan 30:e046142. doi: 10.1161/JAHA.125.046142. Online ahead of print. PMID 41614323
- [Derived] Leatherman SM, Beaudette-Zlatanova B, Robben G, Glassman PA, Woods P, Ferguson RE, Cushman WC, Ishani A. Provider experiences with and attitudes about an embedded pragmatic clinical trial. BMC Prim Care. 2025 Apr 23;26(1):121. doi: 10.1186/s12875-025-02799-w. PMID 40269774
- [Derived] Ishani A, Hau C, Raju S, Wise JK, Glassman PA, Taylor AA, Ferguson RE, Cushman WC, Leatherman SM. Chlorthalidone vs Hydrochlorothiazide and Kidney Outcomes in Patients With Hypertension: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 Dec 2;7(12):e2449576. doi: 10.1001/jamanetworkopen.2024.49576. PMID 39656458
- [Derived] Ishani A, Hau C, Cushman WC, Leatherman SM, Lew RA, Glassman PA, Taylor AA, Ferguson RE. Chlorthalidone vs Hydrochlorothiazide for Hypertension Treatment After Myocardial Infarction or Stroke: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e2411081. doi: 10.1001/jamanetworkopen.2024.11081. PMID 38743423
- [Derived] Klint AL, Leatherman SM, Taylor O, Glassman PA, Ferguson RE, Cushman WC, Ishani A. Telephone informed consent in a pragmatic point-of-care clinical trial embedded in primary care. Contemp Clin Trials. 2023 Aug;131:107239. doi: 10.1016/j.cct.2023.107239. Epub 2023 May 25. PMID 37244366
- [Derived] Raju S, Hau C, Woods P, Flynn M, Sadatis C, McPherson J, Tella A, Ishani A, Ferguson RE, Leatherman SM. Ascertainment of stroke from administrative data to support a pragmatic embedded clinical trial. Contemp Clin Trials. 2023 Jul;130:107214. doi: 10.1016/j.cct.2023.107214. Epub 2023 May 1. PMID 37137378
- [Derived] Leatherman SM, Hau C, Klint A, Glassman PA, Taylor AA, Ferguson RE, Cushman WC, Ishani A. The impact of COVID-19 on a large pragmatic clinical trial embedded in primary care. Contemp Clin Trials. 2023 Jun;129:107179. doi: 10.1016/j.cct.2023.107179. Epub 2023 Apr 7. PMID 37031794

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 72 VA health care systems were enlisted in the trial. A total of 6188 primary care providers were approached for participation in the trial and 4128 (69%) consented. Patients managed by the consented provider were electronically screened for study eligibility. Centralized study recruiters telephoned potential participants and obtained oral informed consent if the patient agreed to participate (n=16595). Of these, 13523 patients were randomized (started participant flow).
Pre-assignment Details: After participants provided verbal informed consent, the patient's provider was sent an electronic order to sign if the provider assented to the patient undergoing study randomization. Provider participation involved agreeing to have their patients approached for trial recruitment by study staff, signing the study drug order, and managing their patient per usual care after randomization. Providers were not randomized.
Period: Overall Study
Arm/Group | Hydrochlorothiazide | Chlorthalidone | Providers
Started | 6767 | 6756 | 4128
Completed | 6312 | 6298 | 4128
Not Completed | 455 | 458 | 0
Not completed — Death | 448 | 446 | 0
Not completed — Withdrawal by Subject | 7 | 12 | 0

BASELINE CHARACTERISTICS:
Population: Analysis and report of baseline information according to the intention-to-treat principle. Baseline characteristics were not collected for providers.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrochlorothiazide | Chlorthalidone | Total
Number analyzed (Participants) | 6767 | 6756 | 13523
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (5.3) | 72.4 (5.4) | 72.4 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211 | 220 | 431
  Male | 6556 | 6536 | 13092
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 257 | 237 | 494
  Not Hispanic or Latino | 6268 | 6281 | 12549
  Unknown or Not Reported | 242 | 238 | 480
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 15 | 28
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1023 | 1004 | 2027
  White | 5225 | 5229 | 10454
  More than one race | 145 | 151 | 296
  Unknown or Not Reported | 361 | 357 | 718
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 79 | 77 | 156
  United States | 6688 | 6679 | 13367
Age [Mean (Standard Deviation); unit: years] | 73.5 (5.3) | 72.4 (5.4) | 72.4 (5.3)
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 31.8 (5.9) | 31.7 (5.8) | 31.8 (5.8)
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 139 (14) | 139 (14) | 139 (14)
Current smoker [Count of Participants; unit: Participants] | 1437 | 1520 | 2957
Resided in rural area [Count of Participants; unit: Participants] | 3079 | 3043 | 6122
History of diabetes [Count of Participants; unit: Participants] | 3062 | 2967 | 6029
History of heart failure [Count of Participants; unit: Participants] | 526 | 525 | 1051
History of myocardial infarction [Count of Participants; unit: Participants] | 258 | 230 | 488
History of stroke [Count of Participants; unit: Participants] | 495 | 534 | 1029
History of myocardial infarction or stroke [Count of Participants; unit: Participants] | 722 | 733 | 1455
Estimated GFR<60 ml/min/1.73 m2 [Count of Participants; unit: Participants] | 1547 | 1550 | 3097
Receiving hydrochlorothiazide at a daily dose of 25 mg [Count of Participants; unit: Participants] — Based on the latest prescription received before study randomization
  Participants | 6402 | 6379 | 12781
Number of antihypertensive drugs prescribed [Mean (Standard Deviation); unit: drugs] — Based on prescriptions received within 182 day before randomization
  drugs | 2.6 (1.0) | 2.6 (1.1) | 2.6 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to Composite Primary Outcome
Description: Time to study primary outcome was defined as years from randomization to the first occurrence of a composite endpoint, consisting of a nonfatal cardiovascular event or non-cancer related death. Nonfatal cardiovascular events included nonfatal myocardial infarction, stroke, hospitalization for heart failure, or urgent coronary revascularization for unstable angina. For participants who had a primary outcome, time to event was determined as the earliest admission or death date. Ascertainment of study outcomes was made with the use of administrative and clinical data obtained from VA EHRs through June 1, 2022, from records of Medicare claims obtained from the Centers for Medicare and Medicaid Services through 2021, and from National Death Index records through 2019. Trial outcomes were ascertained with the use of validated EHR phenotypes and, when needed, manual adjudication. Manually adjudicated outcomes were evaluated by investigators and staff who were unaware of group assignment.
Time Frame: Outcome data collection was performed from study randomization until the participants deceased, withdrawn, or reached end of study (Up to 5.4 years for the first patient enrolled and an average of 2.4 years for all participants).
Population: Analysis of primary outcome was performed according to the intention-to-treat principle.
Measure: Mean (Standard Deviation); unit: Years
Arm/Group | Hydrochlorothiazide | Chlorthalidone
Number analyzed (Participants) | 6767 | 6756
Years | 1.5 (1.0) | 1.5 (1.0)
Statistical Analysis 1: Comparison: Hydrochlorothiazide vs Chlorthalidone; Primary analyses were performed with the use of unadjusted log-rank tests that were stratified according to VA health care system; Test type: Superiority; p = 0.45, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.94 to 1.16]

2. Secondary Outcome: Proportion of Participants Had Nonfatal Myocardial Infarction
Description: Secondary outcomes were the individual components of the primary outcome. Ascertainment of study outcomes was made with the use of administrative and clinical data obtained from VA EHRs through June 1, 2022, from records of Medicare claims obtained from the Centers for Medicare and Medicaid Services through 2021, and from National Death Index records through 2019. Trial outcomes were ascertained with the use of validated EHR phenotypes and, when needed, manual adjudication. Manually adjudicated outcomes were evaluated by investigators and staff who were unaware of group assignment.
Time Frame: as for outcome 1
Population: Analysis of secondary outcome was performed according to the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrochlorothiazide | Chlorthalidone
Number analyzed (Participants) | 6767 | 6756
Participants | 140 | 142

3. Secondary Outcome: Proportion of Participants Had Nonfatal Stroke
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Analysis of secondary outcome was performed according to the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrochlorothiazide | Chlorthalidone
Number analyzed (Participants) | 6767 | 6756
Participants | 83 | 83

4. Secondary Outcome: Proportion of Participants Had Hospitalization for Heart Failure
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Analysis of secondary outcome was performed according to the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrochlorothiazide | Chlorthalidone
Number analyzed (Participants) | 6767 | 6756
Participants | 232 | 242

5. Secondary Outcome: Proportion of Participants Had Unstable Angina Leading to Urgent Coronary Revascularization
Description: as for outcome 2
Time Frame: Collection of outcome data were performed from randomization until participants deceased, withdrawn, or reached end of study (Up to 5.4 years for the first patient enrolled and an average of 2.4 years for all participants).
Population: Analysis of secondary outcome was performed according to the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrochlorothiazide | Chlorthalidone
Number analyzed (Participants) | 6767 | 6756
Participants | 13 | 20

6. Secondary Outcome: Proportion of Participants Deceased and Not Related to Cancer
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Analysis of secondary outcome was performance according to the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrochlorothiazide | Chlorthalidone
Number analyzed (Participants) | 6767 | 6756
Participants | 354 | 359

7. Primary Outcome: Proportion of Participants Had a Composite Primary Outcome
Description: The primary outcome was the first occurrence of a composite endpoint consisting of a nonfatal cardiovascular event or non-cancer related death. Nonfatal cardiovascular events included nonfatal myocardial infarction, stroke, hospitalization for heart failure, or urgent coronary revascularization for unstable angina. Time to the first event was computed based on the earliest hospital admission or death dates. Ascertainment of study outcomes was made with the use of administrative and clinical data obtained from VA EHRs through June 1, 2022, from records of Medicare claims obtained from the Centers for Medicare and Medicaid Services through 2021, and from National Death Index records through 2019. Trial outcomes were ascertained with the use of validated EHR phenotypes and, when needed, manual adjudication. Manually adjudicated outcomes were evaluated by investigators and staff who were unaware of group assignment.
Time Frame: as for outcome 1
Population: Analysis of primary outcome was performed according to the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Hydrochlorothiazide | Chlorthalidone
Number analyzed (Participants) | 6767 | 6756
Participants | 675 | 702

ADVERSE EVENTS:
Time Frame: Safety data collection was performed from study randomization until the participants deceased, withdrawn, or reached end of study (Up to 5.4 years for the first patient enrolled and an average of 2.4 years for all participants).
Description: Adverse events (AE) were collected based on the 21 CFR 312.32, International Conference on Harmonisation (ICH) for Clinical Safety Data Management (ICH-E2A), and Cooperative Studies Program (CSP) Global standard operating procedure definitions. All-cause mortality and hospitalization were monitored and reported as serious adverse events. Expected adverse events of interest were specified in the study protocol and captured from VA electronic medical records. AEs were not collected for providers.
Groups:
- Hydrochlorothiazide: Hydrochlorothiazide daily dose of 50 mg or 25 mg for duration of study
  Hydrochlorothiazide (HCTZ): Thiazide-type diuretic. Daily dose of 50 or 25 mg for duration of the study.
- Chlorthalidone: Chlorthalidone daily dose of 25 mg or 12.5 mg for duration of study
  Chlorthalidone: Thiazide-type diuretic. Daily dose of 25 or 12.5 mg for duration of the study.
Arm/Group | Hydrochlorothiazide | Chlorthalidone
All-Cause Mortality (participants affected / at risk) | 448/6767 | 446/6756
Serious Adverse Events (participants affected / at risk) | 1977/6767 | 1990/6756
Other Adverse Events (participants affected / at risk) | 1229/6767 | 1397/6756
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydrochlorothiazide (N=6767) | Chlorthalidone (N=6756)
All-cause hospitalization (General disorders) | 1826 | 1825
All-cause mortality (General disorders) | 448 | 446
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hydrochlorothiazide (N=6767) | Chlorthalidone (N=6756)
New allergic or adverse reaction to thiazide-type diuretic (General disorders) | 21 | 109
Hypokalemia (General disorders) | 298 | 406
Hyponatremia (General disorders) | 362 | 366
Renal failure (General disorders) | 58 | 61
New onset of diabetes (General disorders) | 240 | 258
Acute gout episode (General disorders) | 100 | 101
Hospitalization for acute kidney injury (General disorders) | 512 | 495

LIMITATIONS AND CAVEATS:
This trial had several important limitations:

* most patients treated with hydrochlorothiazide, including the VA population, received 12.5 to 25 mg, and only 5% in this trial had been receiving 50 mg of hydrochlorothiazide at baseline.
* only a subset of follow-up data from Medicare and NDI were available at the time of reporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-10-26): https://cdn.clinicaltrials.gov/large-docs/17/NCT02185417/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT02185417/SAP_003.pdf
  • Informed Consent Form (2021-02-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT02185417/ICF_004.pdf